CLINICAL TRIAL: NCT00001881
Title: Clinical Manifestations of Mutations in Genes Linked to Familial Cardiomyopathy
Brief Title: Signs and Symptoms of Genetic Abnormalities Linked to Inherited Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990065; 99-H-0065
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Cardiomyopathy, Hypertrophic, Familial
Keywords: Cardiac Hypertrophy; Genetics; Phenotypes; Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic, Familial; Cardiomegaly; Cardiomyopathy, Hypertrophic

SUMMARY:
Genetically inherited heart diseases (familial cardiomyopathies) are conditions affecting the heart passed on to family members through abnormalities in genetic information. These conditions are responsible for many heart related deaths and illnesses.

In this study researchers hope to determine the signs and symptoms (clinical correlation) associated with specific genetic abnormalities causing inherited heart diseases.

In order to do this, researchers plan to evaluate patients and family members of patients diagnosed with inherited heart disease. Patients participating in the study will undergo several tests including blood tests, electrocardiograms (EKG), and echocardiograms. Patients may also be asked to undergo an MRI of the heart to provide a clearer picture of it.

Patients participating in this study may not be directly benefited by it. However, information gathered from the study may contribute to the medical care, treatment, and prevention of problems for others in the future.

DETAILED DESCRIPTION:
Familial cardiomyopathy (FC) often demonstrates both non-allelic and allelic genetic heterogeneity. We propose to determine the clinical correlates of specific genetic defects which cause FC by identifying and expanding a set of kindreds with identical and distinct molecular defects.

ELIGIBILITY:
Individuals with cardiomyopathy referred for evaluation to the NIH.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9999
Dates: Start 1999-03; Study Completion 2001-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fananapazir L, Epstein ND. Prevalence of hypertrophic cardiomyopathy and limitations of screening methods. Circulation. 1995 Aug 15;92(4):700-4. doi: 10.1161/01.cir.92.4.700. No abstract available. PMID 7641346
- [Background] Wigle ED, Rakowski H, Kimball BP, Williams WG. Hypertrophic cardiomyopathy. Clinical spectrum and treatment. Circulation. 1995 Oct 1;92(7):1680-92. doi: 10.1161/01.cir.92.7.1680. PMID 7671349
- [Background] Fananapazir L, McAreavey D. Hypertrophic cardiomyopathy: evaluation and treatment of patients at high risk for sudden death. Pacing Clin Electrophysiol. 1997 Feb;20(2 Pt 2):478-501. doi: 10.1111/j.1540-8159.1997.tb06206.x. PMID 9058851